CLINICAL TRIAL: NCT00911586
Title: Pharmacokinetic Study to Determine Time to Steady-state of an Oral Testosterone Undecanoate Formulation in Hypogonadal Men.
Brief Title: Pharmacokinetic Study to Determine Time to Steady-state
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-09009
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Male Hypogonadism; Primary Hypogonadism; Secondary Hypogonadism
MeSH Terms: conditions — Eunuchism; Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone Undecanoate (Experimental): Oral testosterone undecanoate, 200 mg testosterone (T) as TU, twice daily for 28 days.
  Interventions: Drug: Testosterone undecanoate

INTERVENTIONS:
Drug: Testosterone undecanoate

SUMMARY:
The purpose of the study is to confirm how long (i.e., how many days) it takes to reach steady-state when testosterone undecanoate is administered twice daily.

DETAILED DESCRIPTION:
Serum testosterone levels will be obtained in hypogonadal (serum testosterone <300 ng/dL) males receiving testosterone undecanoate capsules administered twice daily. Serum samples will be obtained consecutively in the morning on several days during one month of open-label treatment to confirm the time at which steady-state is reached.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18-75
* Morning serum testosterone (T) <300 ng/dL on two occasions
* Naive to androgen-replacement therapy or willing to wash-out from current T therapy

Exclusion Criteria:

* Significant intercurrent disease
* Abnormal prostate digital rectal exam, elevated PSA, AUA symptom score >15 or history of prostate cancer.
* Serum transaminases >2 times upper limit of normal
* Serum bilirubin >2.0 mg/dL
* Hematocrit <35% or >50%
* BMI >36
* Untreated, obstructive sleep apnea.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Flippo, MD, Principal Investigator — Alabama Clinical Therapeutics
Locations (1):
- Alabama Clinical Therapeutics, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Yin AY, Htun M, Swerdloff RS, Diaz-Arjonilla M, Dudley RE, Faulkner S, Bross R, Leung A, Baravarian S, Hull L, Longstreth JA, Kulback S, Flippo G, Wang C. Reexamination of pharmacokinetics of oral testosterone undecanoate in hypogonadal men with a new self-emulsifying formulation. J Androl. 2012 Mar-Apr;33(2):190-201. doi: 10.2164/jandrol.111.013169. Epub 2011 Apr 7. PMID 21474786

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Undecanoate: Oral testosterone undecanoate, 200 mg testosterone (T) as TU, twice daily for 28 days.
  Testosterone undecanoate: Oral testosterone undecanoate, 200 mg testosterone (T) as TU, twice daily for 28 days
Period: Overall Study
Arm/Group | Testosterone Undecanoate
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone Undecanoate
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Serum T Concentration at Steady State
Description: Serum T at steady state by evaluating the day-to-day changes in pre-dose concentrations on Days 1, 3, 5, 6, and 7 of treatment.
Time Frame: pre-dose on Days 1, 3, 5, 6, and 7
Population: All participants were included in the analysis population
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Groups:
- Testosterone Undecanoate: Oral testosterone undecanoate, 200 mg testosterone (T) as TU, twice daily for 28 days.
  Testosterone undecanoate
Arm/Group | Testosterone Undecanoate
Number analyzed (Participants) | 15
ng/dL | -4.077 (16.020)
Statistical Analysis 1: Comparison: Testosterone Undecanoate; Test type: Other — Part 1 of piecewise linear regression model; p = 0.8060, Regression, Linear; Part 1 of piecewise linear regression model; Slope = -4.077, Standard Error of Mean 16.020 — Part 1 of piecewise linear regression model

2. Primary Outcome: Serum T Concentration at Steady-State
Description: Serum T at steady-state by evaluating the day-to-day changes in pre-dose concentrations on Days 10, 14, 17, 21, 24, 27, and 28 of treatment.
Time Frame: pre-dose on Days 10, 14, 17, 21, 24, 27, and 28
Population: All participants were included in the analysis population
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | Testosterone Undecanoate
Number analyzed (Participants) | 15
ng/dL | 4.114 (18.456)
Statistical Analysis 1: Comparison: Testosterone Undecanoate; Test type: Other — Part 2 of piecewise linear regression model; p = 0.8286, Regression, Linear; Part 2 of piecewise linear regression model; Slope = 4.114, Standard Error of Mean 18.456 — Part 2 of piecewise linear regression model

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Testosterone Undecanoate
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Undecanoate (N=15)
Belching (Gastrointestinal disorders) | 1 (1)
Gout Flareup (Metabolism and nutrition disorders) | 1 (1)
Irritabililty (General disorders) | 1 (1)
Lower Extremity Edema (General disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Worsening sciatica (Nervous system disorders) | 1 (1)
Stomach bloating (Gastrointestinal disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes